CLINICAL TRIAL: NCT04897542
Title: A Prospective Study to Evaluate the Lesion Detection Ability of Gallium-68 NODAGA-JR11 for the Diagnostic Imaging of Metastatic, Well-differentiated Neuroendocrine Tumors Using PET/CT
Brief Title: Gallium-68 NODAGA-JR11 PECT/CT in Neuroendocrine Tumors
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Weibing Miao, PhD, Director, Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FirstAHFujian8
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients will undergo a Gallium-68 NODAGA-JR11 PET/CT as well as a Gallium-68 DOTATATE PET/CT (Experimental): Each patient receive a single intravenous injection of Gallium-68 DOTATATE (40ug/150-200MBq) PET/CT, and undergo PET/CT scan at 40-60 min post-injection.
  All patients have to do a Gallium-68 NODAGA-JR11 PET/CT scan (40ug/150-200MBq, 40-60 min post-injection) for comparison on the next day of DOTATATE scan.
  Interventions: Drug: Gallium-68 NODAGA-JR11

INTERVENTIONS:
Drug: Gallium-68 NODAGA-JR11 — Each patient receive a single intravenous injection of Gallium-68 NODAGA-JR11 (40ug/150-200MBq) PET/CT, and undergo PET/CT scan at 40-60 min post-injection.

SUMMARY:
NODAGA-JR11 is a novel somatostatin receptor antagonist, while Gallium-68 DOTATATE is a typical somatostatin receptor agonist. This study is to evaluate the lesion detection ability of Gallium-68 NODAGA-JR11 for the diagnostic imaging of metastatic, well-differentiated neuroendocrine tumors using positron emission tomography / computed tomography (PET/CT).

The results will be compared between antagonist Gallium-68 NODAGA-JR11 and agonist Gallium-68 DOTATATE in the same group of patients.

DETAILED DESCRIPTION:
Patients with histologically confirmed metastatic, well-differentiated neuroendocrine tumors will be recruited in this study.

Each patient received an intravenous injection of 68Ga-DOTATATE (40ug/150-200MBq) on the first day and 68Ga-NODAGA-JR11 (40ug/150-200MBq) on the second day. Whole-body PET/CT scans were performed at 40-60 min after injection on the same scanner. Physiologic normal-organ uptake, lesion numbers, and lesion uptake were compared.

ELIGIBILITY:
Inclusion Criteria:

* • Written informed consent.

  * Patients of either gender, aged ≥ 18 years.
  * Histologically confirmed diagnosis of Metastatic, well-differentiated neuroendocrine tumor.
  * A diagnostic computed tomography (CT) or magnetic resonance imaging (MRI) of the tumor region within the previous 6 months prior to dosing day is available.
  * At least 1 measurable lesion based on RECIST v1.1.
  * Blood test results as follows (White blood cell: ≥ 3*10^9/L, Hemoglobin:

    ≥ 8.0 g/dL, Platelets: ≥ 50x10^9/L, Alanine aminotransferase / Aspartate aminotransferase / Alkaline phosphatase: ≤ 5 times upper limit od normal (ULN), Bilirubin: ≤ 3 times ULN)
  * Serum creatinine: within normal limits or < 120 μmol/L for patients aged 60 years or older.
  * Calculated Glomerular filtration rate (GFR) ≥ 45 mL/min.

Exclusion Criteria:

* • Known hypersensitivity to Gallium-68, to NODAGA, to JR11, to TATE or to any of the excipients of Gallium-68 NODAGA-JR11 or Gallium-68 DOTATATE.

  * Presence of active infection at screening or history of serious infection within the previous 6 weeks.
  * Therapeutic use of any somatostatin analog, including long-acting Sandostatin (within 28 days) and short-acting Sandostatin (within 2 days) prior to study imaging. If a patient is on long-acting Sandostatina, then a wash-out phase of 28 days is required before the injection of the study drug. If a patient is on short-acting Sandostatin, then a wash-out phase of 2 days is required before the injection of the study drug.
  * Any neuroendocrine tumor-specific treatment between antagonist and agonist scans.
  * Prior or planned administration of a radiopharmaceutical within 8 half-lives of the radionuclide used on such radiopharmaceutical including at any time during the current study.
  * Pregnant or breast-feeding women.
  * Current history of any malignancy other than neuroendocrine tumor; patients with a secondary tumor in remission of > 5 years can be included.
  * Any mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study, and/or evidence of an uncooperative attitude.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Standard uptake value (SUV) | From right after tracer injection to 2-hours post-injection
  Determination of SUV for detected lesions and discernible organs of 68Ga-NODAGA-JR11 and 68Ga-DOTATATE scan.

SECONDARY OUTCOMES:
Lesion numbers | From right after tracer injection to 2-hours post-injection
  Determination of lesion numbers of 68Ga-NODAGA-JR11 and 68Ga-DOTATATE scan.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian

IPD SHARING:
Plan to Share IPD: No